CLINICAL TRIAL: NCT02113800
Title: Safety and Tolerability of Everolimus as Second-line Treatment in Poorly Differentiated Neuroendocrine Carcinoma / Neuroendocrine Carcinoma G3 (WHO 2010) and Neuroendocrine Tumor G3 - an Investigator Initiated Phase II Study
Acronym: EVINEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Assign Data Management and Biostatistics GmbH (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-NET-0112; CRAD001KDE55T (Other Grant/Funding Number: Novartis); 2012-004550-28 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Poorly Differentiated Malignant Neuroendocrine Carcinoma; Neuroendocrine Carcinoma, Grade 3; Neuroendocrine Carcinoma, Grade 1 [Well-differentiated Neuroendocrine Carcinoma] That Switched to G3; Neuroendocrine Carcinoma, Grade 2 [Moderately Differentiated Neuroendocrine Carcinoma] That Switched to G3; Neuroendocrine Tumor, Grade 3 and Disease Progression as Measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1.)
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Lymphoma, Follicular; Neuroendocrine Tumors | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Patients receive Everolimus orally, 10 mg/day.
  The end of study will be performed when tumor progression has been observed for 28 patients. Patients who are still under treatment at that time may continue with chemotherapy at the discretion of the investigator, but will be excluded from the study.
  Interventions: Drug: Everolimus (Afinitor®)

INTERVENTIONS:
Drug: Everolimus (Afinitor®) — Formulation: 10 mg/day Route: oral (tablet)

SUMMARY:
The study is designed as an open-label, prospective, single arm, multicenter study of everolimus in histologically confirmed, neuroendocrine carcinoma G3 /neuroendocrine tumor G3 after failure of first-line platin-based chemotherapy (open-label pilot study).

The aim of this study is to provide a second line therapy to patients with any type of platinum based first line chemotherapy, to gather data on disease control rate and progression free survival.

DETAILED DESCRIPTION:
As more efficient drugs are urgently needed for the treatment of neuroendocrine tumors the investigator evaluated phosphorylated Mammalian target of rapamycin (mTOR) and effectors in a series of NEC G3 at the Charité Center. Everolimus showed antiproliferative effects in bronchial NET.

In a second approach the data of this study should be the basis to generate another study to further explore everolimus as maintenance therapy in NEC G3/ NET G3.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female ≥ 18 years of age
3. Patients with poorly differentiated neuroendocrine carcinoma, neuroendocrine carcinoma G3 (NEC - G3 according to WHO 2010) or well or moderately differentiated neuroendocrine carcinoma (NET - G1 / G2) that switched to G3 (confirmed by histology) or neuroendocrine tumor G3 (NET G3) and disease progression as measured by RECIST 1.1
4. Progression during or after treatment with first-line platinbased chemotherapy. In NET G3 that switched from NET G2 the line of therapy is determined from the time of revised histology (confirming a G3 NEN)
5. Measurable disease according to RECIST 1.1
6. Performance Status according to Eastern Cooperative Oncology Group (ECOG) status 0 - 2 (Karnofsky Performance status ≥ 80%)
7. Women of child-bearing potential must have a negative pregnancy test
8. Laboratory requirements:

   * Hematology

     * Absolute neutrophil count ≥ 1.5 x 109/L
     * Platelet count ≥ 100 x 10^9/L
     * Leukocyte count ≥ 3.0 x 10^9/L
     * Hemoglobin ≥ 9 g/dL or 5.59 mmol/L
   * Hepatic Function

     * Total bilirubin ≤ 1.5 time the upper limit normal (ULN)
     * Aspartate Aminotransferase (AST) ≤ 3 x ULN in absence of liver metastases, or ≤ 5 x ULN in presence of liver metastases
     * Alanine Aminotransferase (ALT) ≤ 3 x ULN in absence of liver metastases, or ≤ 5 x ULN in presence of liver metastases
   * Renal Function

     * Creatinine clearance ≥ 50 mL/min according to cockroft-Gault formula
   * Metabolic Function

     * Magnesium ≥ lower limit of normal
     * Calcium ≥ lower limit of normal
   * Others:

     * CRP (PCT if CRP is elevated to exclude infection)
     * negative urinary screening test for leukocytes and nitrite (U - stix) to exclude urinary tract infection

Exclusion Criteria:

1. Known or suspected allergy or hypersensitivity reaction to any of the components of study treatment or their excipients.
2. Previous therapy with mTOR inhibitor
3. Radiotherapy :

   * Concurrent radiotherapy involving target lesions used for this study.
   * Concurrent palliative radiation (but radiation for non-target lesions is allowed if other target lesions are available outside the involved field)
   * previous pre-operative or post-operative radiotherapy within 3 months before study treatment
4. History of other malignant tumors within the last 5 years, except basal cell carcinoma or curatively excised cervical carcinoma in situ
5. Known brain metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and steroids
6. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment
7. Inadequate pulmonary function according to the Investigator's judgment, history of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
8. Known active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or HIV infection
9. Serious concomitant disease or medical condition that in the judgment of the investigator renders the patient at high risk from treatment complication
10. Any systemic disease requiring oral intake of corticosteroids (except for replacement therapy of corticosteroids - hydrocortisone in case of adrenal or pituitary insufficiency)
11. Hearing loss ≥ Grade 3 (CTCAE v4.03)
12. Patient pregnant or breast feeding, or planning to become pregnant within 8 weeks after the end of treatment
13. Patient (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 8 weeks (male or female) after the end of treatment.
14. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 28 days prior to treatment start
15. Concurrent treatment with inhibitors (e.g. itraconazole, ketoconazole) and inducers (e.g. phenytoin, rifampicin) of Cytochrome P450 3A4 (CYP3A4) and / or the multidrug efflux pump P-glycoprotein (PgP).
16. Known drug abuse/alcohol abuse
17. Peripheral polyneuropathy ≥ Grade 2 (CTCAE v4.03)
18. Active chronic inflammatory bowel disease
19. Any condition which might interfere with study objectives (e.g. infections) or would limit the patient's ability to complete the study in the opinion of the investigator
20. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities. (AMG §40, Abs. 1 No. 4)
21. Affected persons who might be dependent on the sponsor or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | approx. 18 month
  Incidence of adverse events (AEs) overall and by severity, and serious adverse events (SAEs). Severity will be assessed using the National Cancer Institute-Common Toxicity Criteria (NCI-CTC) for Adverse Events, version 4.03 (CTCAEv4.03).
  To evaluate tolerability and safety of everolimus in second-line treatment of poorly differentiated neuroendocrine carcinoma / neuroendocrine carcinoma G3 according to WHO 2010 and neuroendocrine tumors G3.

SECONDARY OUTCOMES:
Progression free survival (PFS) | approx. 18 month
  Progression free survival (PFS) as the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse as per local radiology assessment using Response Evaluation Criteria in Solid Tumors (RECIST 1.1.)
Objective response rate (ORR) | approx. 18 month
  Objective response rate defined as the rate of best overall response (CR+PR), determined by RECIST V 1.1.
Disease control rate (DCR) | approx. 18 month
  Disease control rate defined as the rate of best overall response and stable disease (CR+PR+SD), determined by RECIST V 1.1.
Duration of response (DR) | approx. 18 month
  Duration of response is defined as the time from onset of the first objective tumor response (CR/PR) to objective tumor progression or death from any cause.
Overall Survival (OS) | approx. 18 month
  OS is defined as the time from date of randomization to the date of death from any cause. If a patient is not known to have died at the date of analysis cut-off, the OS will be censored at the last date of contact.
Quality of life | approx. 18 month
  Quality of life (HRQoL) will be evaluated using the European Organisation for Research and Treatment of Cancer (EORTC), to assess the quality of life of cancer patients questionnaire (QLQ-C30)
chromogranin A & B | approx. 12 month
  Percentage of patients showing normalization or a decrease of chromogranin A & B
Time to Progression (TTP) | approx. 18 month
  Time to progression (TTP) is the time from date of start of treatment to the date of event defined as the first documented progression due to underlying cancer.
neuron-specific enolase | approx. 12 month
  Percentage of patients showing normalization or a decrease of neuron-specific enolase
progastrin releasing peptide | approx. 12 month
  Percentage of patients showing normalization or a decrease of progastrin releasing peptide.
Correlation mTOR pathway components in tumor tissue to tumor response | approx. 18 month
  To explore expression of mTOR pathway components in tumor tissue (archive) in correlation to tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Pavel, Prof. Dr., Principal Investigator — Charité-Universitätsmedizin
Locations (1):
- Charité-Universitätsmedizin, Medizinische Klinik m. S. Hepatologie und Gastroenterologie, Campus Virchow-Klinikum, Berlin, Germany

REFERENCES:
- [Derived] Jungels C, Deleporte A. State of the art and future directions in the systemic treatment of neuroendocrine neoplasms. Curr Opin Oncol. 2021 Jul 1;33(4):378-385. doi: 10.1097/CCO.0000000000000740. PMID 33973550
- See also: Working Group for Medical Oncology (AIO) from the German Cancer Society (DKG) — http://www.aio-portal.de